CLINICAL TRIAL: NCT05648097
Title: Baldachin-Study: Ceiling HEPA-filtration to Prevent Nosocomial Transmission of COVID-19 in Open-space Multiple Bed Patient Areas
Brief Title: Baldachin: Ceiling HEPA-filtration to Prevent Nosocomial Transmission of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Balda01
Record Dates: First submitted 2022-12-12; First posted 2022-12-13 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: Sars-CoV2; Aerosols; Infection transmission; Infection risk; Respiratory Tract Infections; Virus Diseases
MeSH Terms: conditions — COVID-19; Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients exposed to a patient with COVID-19 isolated at the site - standard of care
- Baldachin-Intervention (Active Comparator): Patients exposed to a patient with COVID-19 isolated at the site - under Baldachin
  Interventions: Device: Baldachin

INTERVENTIONS:
Device: Baldachin — Environmental intervention: Equipment of a patient space of a patient with confirmed COVID-19 in open-space multiple bed Intermediate Care Unit areas with a mobile, optimally placed high efficiency particulate air ("HEPA")-equivalent air filtration unit ("Baldachin") in addition to existing room ventilation and hospital policy infection prevention and control measures.
  Arms: Baldachin-Intervention

SUMMARY:
In this study, a patient space occupied by a patient with confirmed COVID-19 in an open-space multiple bed area in the Intermediate Care Unit will be equipped with a mobile, optimally placed high efficiency particulate air ("HEPA")-equivalent air filtration unit ("Baldachin") in addition to existing hospital policy infection prevention and control measures. The investigators are going to evaluate this intervention regarding its capacity to prevent the nosocomial onwards transmission of Sars-COV2 to patients located in the same multiple-bed open space patient area.

DETAILED DESCRIPTION:
SARS-CoV-2 transmission includes a considerable amount of long-distance aerosol transmission. Ideal isolation is in single rooms. Isolation in special care multiple bed open-space patient areas (e.g. in the Intensive and Intermediate Care Unit) is set back to onsite isolation with distancing and ventilation as partial mitigation measures against nosocomial transmission.

The investigators want to assess the effect of supplementation of existing room ventilation by means of an optimally placed mobile high efficiency particulate air ("HEPA") filtration unit ("Baldachin") in the ceiling area over confirmed COVID-19 infected patients on nosocomial onwards transmission to patients located in the same open-space multiple bed area. In order to quantify the effect, the investigators will determine the proportion of nosocomially infected individuals as assessed by nasopharyngeal swab on day 4 after the last exposure amongst all in the same room exposed patients in cardiovascular open-space Intermediate Care Unit rooms with "Baldachin" vs. open-space Intermediate Care Unit rooms without "Baldachin".

ELIGIBILITY:
Inclusion Criteria:

* Adult inpatients of included open-space IMC units with lab-confirmed SARS-CoV-2 infection, symptom onset or date of test ≤10 days prior inclusion.

Exclusion Criteria:

* Pregnancy, unability to give consent (e.g. informed consent form not available in patient language or non-judicious)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of nosocomially infected individuals within 4 days after exposure | 4 days after last exposure
  Assessed by nasopharyngeal swab on day 4 after the last exposure amongst all in the same room exposed patients in cardiovascular open-space Intermediate Care Unit ("IMC") rooms with the environmental interventions vs. open-space IMC rooms without the environmental intervention

SECONDARY OUTCOMES:
Exposure duration | Period when exposed to a patient with confirmed COVID-19 in the same room
  Expected to be on average hours up to a few days
Proportion of immunocompromised patients among those exposed | At the time of exposure
  e.g. patients under treatment with steroids, chemotherapy
Preexisting air change rate per hour in the rooms where exposure occurs | At the time of exposure
Age of exposed patients | At the time of exposure
  As part of the demographic characteristics
Gender of exposed patients | At the time of exposure
  As part of the demographic characteristics
Proportion of nosocomially infected patients within 10 days after exposure | 10 days after last exposure
  As documented in the electronic patient record

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Jent, MD, Principal Investigator — Department of Infectious Diseases Inselspital Bern University Hospital
Locations (1):
- Inselspital Bern University Hospital, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No